CLINICAL TRIAL: NCT00608361
Title: Phase I Pharmacokinetic Study of Dasatinib (BMS-354825) (NSC-732517) in Patients With Advanced Malignancies and Varying Levels of Liver Dysfunction
Brief Title: Dasatinib in Treating Patients With Solid Tumors or Lymphomas That Are Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00792; NCI-2009-00792 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000583976; SWOG-S0711; S0711 (Other: SWOG); S0711 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2008-01-30; First posted 2008-02-06 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Adult B Acute Lymphoblastic Leukemia; Adult Hepatocellular Carcinoma; Adult Nasal Type Extranodal NK/T-Cell Lymphoma; Adult Solid Neoplasm; Adult T Acute Lymphoblastic Leukemia; Advanced Adult Hepatocellular Carcinoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-Cell Lymphoma; Chronic Lymphocytic Leukemia; Cutaneous B-Cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone Lymphoma of Mucosa-Associated Lymphoid Tissue; Hepatosplenic T-Cell Lymphoma; Intraocular Lymphoma; Localized Non-Resectable Adult Liver Carcinoma; Localized Resectable Adult Liver Carcinoma; Lymphomatous Involvement of Non-Cutaneous Extranodal Site; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Nodal Marginal Zone Lymphoma; Progressive Hairy Cell Leukemia Initial Treatment; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Lymphoma; Recurrent Adult Liver Carcinoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-Cell Leukemia/Lymphoma; Recurrent Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides and Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestinal Lymphoma; Splenic Marginal Zone Lymphoma; Stage II Small Lymphocytic Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-Cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IIIA Mycosis Fungoides and Sezary Syndrome; Stage IIIB Mycosis Fungoides and Sezary Syndrome; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-Cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Stage IVA Mycosis Fungoides and Sezary Syndrome; Stage IVB Mycosis Fungoides and Sezary Syndrome; T-Cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Hairy Cell Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Burkitt Lymphoma; Carcinoma, Hepatocellular; Lymphoma, Extranodal NK-T-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Intraocular Lymphoma; Lymphoma, T-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (dasatinib) (Experimental): Patients receive dasatinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of dasatinib in treating patients with solid tumors or lymphomas that are metastatic or cannot be removed by surgery. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of dasatinib in patients with varying degrees of hepatic impairment.

II. To estimate the pharmacokinetic (PK) profile of this drug in patients with varying degrees of hepatic impairment.

III. To assess the safety profile and dose-limiting toxicities (if any) of dasatinib in patients with varying degrees of hepatic impairment.

SECONDARY OBJECTIVES:

I. To describe any antitumor efficacy associated with dasatinib administration in patients with varying degrees of hepatic impairment.

II. To examine whether the pharmacokinetic clearance of dasatinib correlates with hepatic function as assessed by Child-Pugh Criteria, the National Cancer Institute (NCI) Organ Dysfunction Working Group Criteria, or other assessments of liver function.

OUTLINE: This is a dose-escalation study.

Patients receive dasatinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed solid tumor or lymphoma that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; patients with a liver mass, elevated alpha-fetoprotein level (>= 500 ng/mL) and positive serology for viral hepatitis, consistent with a diagnosis of hepatocellular carcinoma will be eligible without the need for pathologic confirmation of the diagnosis; all solid and lymphoma tumor types are eligible
* Patients must have measurable or non-measurable disease; x-rays and/or scans for disease assessment must have been completed within 28 days (for measurable disease) or 42 days (for non-measurable disease) prior to registration; all disease must be assessed and documented on the web-based Baseline Tumor Assessment Form
* Patients with brain metastases who require corticosteroids must be on stable or decreasing dose of corticosteroids; patients with known brain metastases must have had brain irradiation (whole brain or gamma knife); patients with untreated (non-irradiated) brain metastases are not eligible; patients on enzyme-inducing anticonvulsant medications (e.g. phenobarbital, phenytoin or carbamazepine) are not eligible
* Patients must not be taking H2-receptor antagonists such as cimetidine, ranitidine, and famotidine, or any proton pump inhibitors, such as omeprazole, lansoprazole, esomeprazole, and pantoprazole; patients must stop these medications within 7 days prior to starting treatment
* Patients must not have had anticancer therapy including chemotherapy, radiotherapy, immunotherapy, or investigational agent within 4 weeks prior to registration, except for targeted agents with half-life known to be < 24 hours; patients must not have had targeted agents with half-life < 24 hours within 2 weeks prior to registration; patients also must have recovered from serious adverse events due to agents administered within these acceptable time frames
* Patients must not be planning to receive concurrent radiation, other chemotherapy, immune therapy or any other investigational agents for malignancy while receiving protocol treatment; hormonal treatment for prostate carcinoma may be continued and bisphosphonate treatment for bone disease is permitted
* Patient must not have received prior therapy with dasatinib (BMS-354825)
* Patients for whom there is a strong suspicion of being allergic to dasatinib because of a history of allergic reactions to similar compounds are not eligible
* Patients must not have had major surgical procedures within the last 4 weeks prior to the first planned dose of study drug
* Patients must not be taking therapeutic doses of anticoagulants; low dose warfarin for port prophylaxis is permitted
* Zubrod performance status of 0-2
* Patients may not have any clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged corrected QT interval (QTc) >= 480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients with any cardiopulmonary symptoms of unknown cause (e.g. shortness of breath, chest pain, etc.) should be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation; the patient may be referred to a cardiologist at the discretion of the principal investigator; patients with underlying cardiopulmonary dysfunction should be excluded from the study
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Magnesium >= lower limit of normal (LLN)
* Potassium >= LLN
* Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance >= 60 mL/min/1.73 m^2; if less than the normal range, supplementation should be initiated in the manner deemed appropriate by the treating physician
* Patients with abnormal liver function are eligible and will be grouped according to the criteria; no distinction will be made between liver dysfunction due to metastases and liver dysfunction due to other causes; for patient registration, liver function tests (total bilirubin, aspartate aminotransferase [AST]/alanine aminotransferase [ALT], prothrombin time [PT]/international normalized ratio [INR] and partial thromboplastin time [PTT], and alkaline phosphatase) must be performed within 14 days prior to registration; for patient stratification, liver function tests must be performed within 72 hours of anticipated starting time of protocol treatment; patients must be stratified and treated based on the liver function tests performed within 72 hours prior to treatment; the South West Oncology Group (SWOG) Data Operations Center must be notified in writing in cases where the patient's cycle 1 pre-treatment liver function tests result in stratification to a dysfunction group different from how the patient was classified at registration
* Patients with biliary obstruction for which a shunt has been placed are eligible, provided the liver function tests have stabilized (two measurements at least two days apart that put the patient in the same hepatic dysfunction stratum will be accepted as evidence of stable hepatic function); there must be no evidence of biliary sepsis and at least 2 weeks must have elapsed after the placement of a biliary shunt
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; since interaction with dasatinib and oral contraceptives is possible, a barrier method should be used and oral contraceptives are not permitted; a negative pregnancy test is required within 72 hours prior to starting therapy for women of reproductive potential; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients who have experienced any of the following within the 12 months prior to starting protocol treatment are not eligible: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or significant pulmonary embolus
* Patients with ongoing cardiac dysrhythmias of NCI Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2, atrial fibrillation of any grade, or QTc interval > 470 msec for females or > 450 msec for males are not eligible
* Patients with baseline pleural effusion are not eligible
* Patients must not have active gastrointestinal bleeding
* Patients with the inability to take oral medications, with a diagnosis of malabsorption syndromes or with significant bowel resection affecting absorption are not eligible
* Patients with a clinically significant pleural effusion/ fluid retention/pericardial effusion are not eligible; patients with a history of pleurodesis and previous pleural effusion (malignant or non-malignant) may be eligible but treated with caution; patients with previous history of ascites may be treated
* Patients with uncontrolled serious intercurrent medical illness including, but not limited to ongoing or serious active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia, uncontrolled diarrhea or psychiatric illness/social situations that would limit compliance with study requirements are not eligible
* Patients known to be human immunodeficiency virus (HIV)-positive are not eligible; however, patients will not routinely be screened for HIV
* Patients must be willing to undergo pharmacokinetic sampling
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and identification (ID) number must be provided to the Statistical Center in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the data base

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of dasatinib, defined as the highest dose level at which less than 33% of 6-9 evaluable patients experience dose-limiting toxicity | 28 days
  Toxicity will be graded according to the NCI CTCAE v3.0.
Pharmacokinetic parameters of dasatinib | Days 1 and 8 of course 1
  Area under curve (AUC)(to infinity), AUC(to 24 hours), and maximum concentration (Cmax) analyzed in the natural log scale. For each PK parameter, the mean difference between the recommended dose for a liver impairment group and the normal liver function group dosed at 140 mg OD (equivalent to ratios of geometric means in the non-log scale) will be tested against 0 at a one-sided 0.05 significance level to detect an increase in the liver impairment group (equivalent to a 2-sided 90% confidence interval).

OTHER OUTCOMES:
Liver dysfunction data | Baseline
  The Child-Pugh classification (CPC), NCI Organ Dysfunction Working Group (ODWG) Stratification Criteria for all patients will be collected at baseline and correlated to the toxicities and pharmacokinetic data seen with dasatinib in an exploratory analysis. Clearance estimates for each liver impairment group based upon the NCI ODWG Criteria, CPC Scheme, will be correlated with drug clearance. Ultimately, the predictive value of these various different methods of grouping organ dysfunction patients will be compared to determine if any method is better able to predict dasatinib clearance.

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, Principal Investigator — SWOG Cancer Research Network
Locations (23):
- United States (23):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Henry Ford Hospital, Detroit, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Audie L Murphy Veterans Affairs Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington